CLINICAL TRIAL: NCT02758730
Title: A Randomized, Placebo-controlled, Parallel Group, Patient-blind, Single-center Phase I Pilot Study Assessing Tolerability and Safety and Exploring the Immunogenicity and Therapeutic Activity of AFFITOPE® PD01A, a New Vaccine Against Alpha-synuclein, in Patients With PD-GBA
Brief Title: Study Assessing Tolerability and Safety and Exploring the Immunogenicity and Therapeutic Activity of AFFITOPE® PD01A in PD-GBA Patients
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Affiris AG (Industry)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AFF010; 2016-001462-28 (EudraCT Number)
Record Dates: First submitted 2016-04-26; First posted 2016-05-02 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Parkinson's Disease
Keywords: GBA mutation
MeSH Terms: conditions — Parkinson Disease | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AFFITOPE® PD01A + Adjuvant (Experimental): 3 injections of 75µg AFFITOPE® PD01A/ adjuvanted, once every 4 weeks
  Interventions: Biological: AFFITOPE® PD01A + Adjuvant
- Adjuvant without active component (Placebo Comparator): 3 injections of Placebo once every 4 weeks
  Interventions: Biological: Adjuvant without active component

INTERVENTIONS:
Biological: AFFITOPE® PD01A + Adjuvant — s.c. injection
  Arms: AFFITOPE® PD01A + Adjuvant
Biological: Adjuvant without active component — s.c. injection
  Arms: Adjuvant without active component

SUMMARY:
This is a randomized, placebo-controlled, parallel group, patient-blind, single-center phase I clinical trial of repeated once every 4 weeks administration by subcutaneous injection of AFFITOPE® PD01A, adsorbed to aluminium oxide in 30 patients with PD-GBA over a treatment period of 8 weeks. Patients will be randomized in a 2:1 ratio to two different treatment groups: A) 75 µg AFFITOPE® PD01A, adsorbed to aluminium oxide and B) placebo (= 1 mg aluminium oxide).

Over a study duration of 52 weeks, each patient will receive 3 injections of AFFITOPE® PD01A or placebo during the participation in the clinical trial. Patients will either receive 75 µg AFFITOPE® PD01A adsorbed to 1 mg aluminium oxide or placebo (=1mg aluminium oxide). The treatment group consists of 20 PDGBA patients, the placebo group of 10 PDGBA patients. Male and female patients aged 40 to 80 years can participate in the trial.

AFF010 is part of the project MULTISYN funded by the European Commission (FP7-HEALTH-2013-INNOVATION-1 project; N° HEALTH-F4-2013-602646).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Parkinson's disease and confirmed carrier status for a heterozygous GBA mutation (PDGBA)
* Individuals who present in Hoehn&Yahr Stages I/II/III and fulfill the United Kingdom Parkinson's Disease Society Brain Bank Criteria
* Confirmed carrier status for a heterozygous GBA mutation (PDGBA)-The result of the MRI scan of the patient's brain has to be consistent with the diagnosis of PD
* Written informed consent signed and dated by the patient and, preferentially, the caregiver (caregiver is not mandatory)
* Age between 40 and 80
* In the investigator's opinion, does not have visual or auditory impairments that would reduce the patients' ability to complete study questionnaires or be unable to receive instructions for these
* Female patients of childbearing potential are eligible if they use a medically accepted contraceptive method
* A potential participant treated with conventional PD therapies must be on stable doses for at least 3 months prior to Visit 1 and during the entire trial period
* Accepted PD medications include the following: levodopa (alone or in combination with benserazide, carbidopa), catechol-O-methyltransferase (COMT) inhibitors (entacapone, tolcapone), amantadine, non-ergot dopamine agonists (pramipexol, ropinirol, rotigotine), monoamine oxidase-B (MAO-B) inhibitors (rasagiline, selegiline) and anticholinergic medication
* A potential participant should be on stable doses of all medications he/she is taking because of consisting illnesses according to medical history (except PD therapies, these will be recorded separately) for at least 30 days prior to Visit 1 if considered relevant by the investigator
* Able to communicate well with the investigator, to understand and comply with the requirements of the study

Exclusion Criteria:

* Pregnant women
* Sexually active women of childbearing potential who are not using a medically accepted birth control method
* Participation in another clinical trial within 3 months before Visit 1
* History of questionable compliance to visit schedule; patients not expected to complete the clinical trial
* Presence or history of allergy to components of the vaccine if considered relevant by the investigator
* Contraindication for MRI imaging such as metallic implants (e.g. endoprosthesis, stents, cardiac pacemakers) which are not MR compatible at 3.0 Tesla with the given MR protocol, other foreign metal bodies (e.g. bullets, metal splinters, e.g.) or claustrophobia
* Missing agreement to be informed about incident findings and consultation of a neuroradiologist
* Contraindication for PET, that is, pregnancy and breast feeding.
* Ongoing participation in other interventional studies or clinical trials using radiotracers
* Dementia according to Diagnostic and Statistical Manual (DSM) IV criteria
* History and/or presence of autoimmune disease, if considered relevant by the investigator
* Recent (≤3 years since last specific treatment) history of cancer (Exceptions: non-melanoma skin cancer, intraepithelial cervical neoplasia)
* Active infectious disease (e.g., Hepatitis B, C)
* Presence and/or history of Immunodeficiency (e.g., HIV)
* Significant systemic illness (e.g., chronic renal failure, chronic liver disease, poorly controlled diabetes, poorly controlled congestive heart failure, other deficiencies), if considered relevant by the investigator
* History of significant psychiatric illness such as schizophrenia, bipolar affective disorder or psychotic depression
* Parkinson-like disease secondary to drug therapy side effects (e.g., due to exposure to medications that deplete dopamine [reserpine, tetrabenazine] or block dopamine receptors [neuroleptics, antiemetics])
* Parkinson-plus syndromes (e.g., multiple system atrophy (MSA), progressive supranuclear palsy (PSP)), Dementia with Lewy Bodies (DLB)
* Heredodegenerative disorders other than PDGBA, evidence for other genetic forms of PD (e.g. LRRK2, Parkin gene mutations)
* Alcoholism or substance abuse within the past year (alcohol or drug intoxication)
* Prior and/or current treatment with experimental immunotherapeutics including Intravenous Immunoglobulin (IVIG)
* Prior and/or current treatment with immune modulating drugs:

  1. Interleukins, Interferons, Tumor Necrosis Factor (TNF) and analogues, colony stimulating factor compounds
  2. Ciclosporin, Tacrolimus, Sirolimus and analogues
  3. Cytostatic drugs and certain DMARD for rheumatoid arthritis (and similar autoimmune disorders) (e.g. Cyclophosphamid, Azathioprin, methotrexate, sulfasalazine, leflunomide, sodium aurothiomalate (Gold), cyclosporin) and analogues
  4. Systemic (gluco)corticoid therapy
  5. All antibody therapies (e.g., anti cluster of differentiation 3 (CD3), anti cluster of differentiation 25 (CD25) or also anti-lymphocyte globulins) that might modulate, enhance or weaken an immune response
* Change in dose of standard treatments for PD within 3 months prior to Visit 1
* Change in dose of previous and current medications which the patient is taking because of consisting illnesses according medical history (except PD therapies, these will be recorded separately) within the last 30 days prior to Visit 1, if clinically relevant
* Treatment with deep brain stimulation
* Venous status rendering it impossible to place an i.v. access

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients who withdraw due to Adverse Events (AEs) and reason for withdrawal | 52 weeks
Occurrence of any Serious Adverse Event (SAE) possibly, probably or definitely related to the study vaccine at any time during the study | 52 weeks
Occurrence of any Grade 3 or higher AEs possibly, probably or definitely related to the study vaccine within 4 weeks after the vaccinations | 12 weeks (week 0 to 12)
Occurrence of solicited local AEs | up to 52 weeks
  Injection site pain, erythema (redness), hyperthermia at injection site, itching, edema (swelling), induration [hardening], granuloma within 1 week (Day 1-7) after the vaccinations: Severity and duration
Occurrence of solicited systemic AEs | up to 52 weeks
  Headache, myalgia (muscle pain), fever, fatigue, nausea within 1 week (Day 1-7) after the vaccinations: Severity and duration.
Occurrence of unsolicited non-serious AEs within four weeks after the vaccinations | 12 weeks (week 0 to 12)
  Severity, duration and relationship to vaccination

SECONDARY OUTCOMES:
Immunological activity of AFFITOPE® vaccine PD01A over time (study period) | 52 weeks
  Titer of immunoglobulin G (IgG) Abs specific for the immunizing peptide (PD01A), the carrier (KLH) and the target (targeted native α-Synuclein (aSyn) epitope coupled to bovine serum albumin (BSA) (mandatory) or presented in different forms - particularly monomers, pre-fibrils and fibrils (optional)) assessed by Enzyme-Linked Immunosorbent Assay (ELlSA) (or an equivalent method)
Imaging efficacy variables at visit 6 (or EDV) compared to baseline | 52 weeks
  11C-Pittsburgh Compound B (11C-PIB), 18F-Fluorodeoxyglucose-Positron Emission Tomography (18F-FDG-PET), resting-state functional magnetic resonance imaging (fMRI), diffusion-weighted/tensor magnetic resonance imaging (MRI), Magnetic Resonance-Spectroscopy
Biomarker data at visit 6 (or EDV) compared to baseline | 52 weeks
  β-Glucocerebrosidase (GCase) enzyme activity

OTHER OUTCOMES:
Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) I, II, III and IV at visit 5 and visit 6 (or EDV) compared to baseline | 52 weeks
  Change in motor/non-motor symptoms over time
Parkinson's Disease Quality of Life-39 (PDQ-39) at visit 5 and visit 6 (or EDV) compared to baseline | 52 weeks
  Change in non-motor PD symptoms over time
Investigator's global evaluation scale at visit 5 and visit 6 (or EDV) | 52 weeks
  Change in motor PD symptoms over time. The overall change in the severity of patient's illness, compared to patient's condition at the start of this clinical trial (Visit 1).
Cognitive scales at visit 5 and visit 6 (or EDV) compared to baseline | 52 weeks
  Change in non-motor PD symptoms over time (MOCA, Trail Making Test (TMF) A and B)
Geriatric Depression Scale at visit 5 and visit 6 (or EDV) compared to baseline | 52 weeks
  Change in non-motor PD symptoms over time

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Gasser, Prof. Dr., Principal Investigator — University Hospital Tübingen, 72076 Tübingen, Germany
Locations (1):
- University Hospital Tübingen, Tübingen, Germany